CLINICAL TRIAL: NCT01460732
Title: Home Versus Ambulatory Monitoring in the Assessment of the Diurnal Blood Pressure Profile and the Detection of Non-Dippers
Brief Title: Home Versus Ambulatory Monitoring, Diurnal Blood Pressure Profile, Detection of Non-Dippers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NOCTURNAL
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension
Keywords: Hypertension; Nocturnal BP dipping; Home Blood pressure Monitoring; Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Other): All eligible patients in the study consist a single group and the same intervention is assigned to all of them.
  Interventions: Device: Blood Pressure Monitoring

INTERVENTIONS:
Device: Blood Pressure Monitoring — Home Blood pressure Monitoring Nocturnal-Home Blood Pressure Monitoring Ambulatory Blood Pressure Monitoring
  Other Names: Microlife WatchBP Home Nocturnal; Microlife WatchBP O3

SUMMARY:
This is a cross-sectional study, including adults, either untreated for hypertension, or under stable treatment for more than four weeks. Assessment will include:

Clinic blood pressure measurements with an automated oscillometric device, 24-hour ambulatory blood pressure monitoring Home blood pressure monitoring during morning, evening and nocturnal measurements with the same device.

DETAILED DESCRIPTION:
Eligible patients, as described in Inclusion/Exclusion Criteria, will be instructed to use Microlife WatchBP Home-Nocturnal oscillometric device, in order to measure their BP two times with one-minute interval, in the morning between 6 and 9 am and in the evening between 6 and 9 pm respectively for six days. These six days shall be normal working days, selected be the patient, within a time-frame of two weeks approximately. Patients should be sitting for at least five minutes and calm. During three out of those six days, they will apply and activate the same device, in order to take BP measurements while they will be asleep. Those measurements are going to be taken automatically by the device, the first 2-hours after the activation and another two with one-hour interval. Measurements will be averaged as awake and asleep BP values, with a potential to derive, if so wished, separate averages of awake-morning and awake-evening BP values.

Microlife WatchBP O3 Ambulatory Blood Pressure Measurement (ABPM) device will be applied by a doctor to each patient and it will be removed the next day by a doctor. BP measurements will be performed every 20 minutes for 24 hours. BP measurements taken during awake and asleep hours for each patient, will be analyzed separately.

Additionally, triplicate sitting Clinic Blood Pressure measurements, with one-minute interval, will be performed with the Microlife WatchBP Home-Nocturnal device during each patient's visit at the Hypertension Center. Patients will visit Hypertension Center three times, one to apply the ABPM device and one to remove it and provide the Microlife WatchBP Home-Nocturnal device and another one to bring it back. This will take approximately two weeks.

ELIGIBILITY:
Inclusion Criteria:ma

* Patients referred for high blood pressure
* Age over 30 years
* Untreated for hypertension or under stable treatment for 4 weeks or more
* Patients physically and mentally capable for self-measurement of blood pressure at home
* Written informed consent to participate in the study

Exclusion Criteria:

* Sustained arrythmia
* Pregnancy
* Symptomatic cardiovascular disease
* Any other serious disease (renal failure, heart failure, malignancy)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sotiria General Hospital, Athens, Greece

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients analyzed
Period: Overall Study
Arm/Group | All Patients
Started | 81
Completed | 81
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 43
Region of Enrollment [Number; unit: participants]
  Greece | 81

OUTCOME MEASURES:

1. Primary Outcome: Awake Systolic Home Blood Pressure Measurement
Description: Awake Home Blood Pressure measurement includes duplicate BP measurements in the morning and in the evening, as per protocol.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 131.5 (11.2)

2. Primary Outcome: Awake Diastolic Home Blood Pressure Measurement
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 79.9 (7.8)

3. Primary Outcome: Asleep Systolic Home Blood Pressure Measurement
Description: Home Blood Pressure measurement device was applied by the patient himself, in order to perform BP measurements during sleep, as per protocol.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 114.8 (12.2)

4. Primary Outcome: Asleep Diastolic Home Blood Pressure Measurement
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 66.6 (7.9)

5. Primary Outcome: Awake Systolic Ambulatory Blood Pressure Measurement
Description: An Ambulatory Blood Pressure Measurement device is applied by a doctor to each patient for 24 hours and next day it is removed. Measurements taken during patient's awake and asleep hours are analyzed separately.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 130.0 (11.6)

6. Primary Outcome: Awake Diastolic Ambulatory Blood Pressure Measurement
Description: as for outcome 5
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 81.0 (7.6)

7. Primary Outcome: Asleep Systolic Ambulatory Blood Pressure Measurement
Description: as for outcome 5
Time Frame: 2weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 115.2 (10.7)

8. Primary Outcome: Asleep Diastolic Ambulatory Blood Pressure Measurement
Description: as for outcome 5
Time Frame: 2weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 81
mmHg | 67.6 (6.9)

9. Secondary Outcome: Dippers Defined by ABPM and HBPM-Nocturnal
Description: As Dippers are defined the patients who displayed a nocturnal fall (Daytime-Nighttime BP/Daytime BP) in Systolic and/or Diastolic Blood Pressure by 10% or more, by each method. The rest of patients, with a nocturnal fall by less than 10% or even a rise of BP, are consequently defined as Non-Dippers.
Time Frame: 2 weeks
Population: All patients who had their Daytime and Nocturnal BP assessed by both methods.
Measure: Number; unit: percentage of patients
Groups:
- ABPM: Dippers defined by ABPM.
- HBPM-Nocturnal: Dippers defined by HBPM-Nocturnal.
Arm/Group | ABPM | HBPM-Nocturnal
Number analyzed (Participants) | 81 | 81
percentage of patients | 84 | 78

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No